CLINICAL TRIAL: NCT05991791
Title: Adapted and Individualized Intelligent Robotic Interactions to the Ability Spectrum of Children With Autism Spectrum Disorder
Brief Title: Intelligent Robotic Interactions for Children With Autism Spectrum Disorders
Acronym: I-ROBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL23_0056
Record Dates: First submitted 2023-07-28; First posted 2023-08-15 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; children; interventional care; robotics; telepresence
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with autism spectrum disorders (Other)
  Interventions: Other: Early Start Denver Model (ESDM)

INTERVENTIONS:
Other: Early Start Denver Model (ESDM) — Phase A
  * 4 individual sessions (1 per week)
  * Additional time of 15 minutes to evaluate 3 selected tasks of the ESDM
  * Satisfaction Evaluation - Parent
  * Satisfaction Evaluation - Therapist
  Phase B :
  * 11 sessions (1 per week)
  * Additional time of 15 minutes to evaluate 3 selected tasks of the ESDM with the help of the robot Pepper
  * Satisfaction Evaluation - Parent
  * Satisfaction Evaluation - Therapist
  Phase C :
  * 4 sessions (1 per week)
  * Additional time of 15 minutes to evaluate 3 selected tasks of the ESDM without the help of the robot Pepper
  * Satisfaction Evaluation - Parent
  * Satisfaction Evaluation - Therapist
  * All sessions will also be filmed and recorded

SUMMARY:
For several years, studies have been developed on the contribution of social robots as a tool for interventions for children with autism spectrum disorders (ASD). One of the recommended intervention models is the ESDM (Early Start Denver Model). It consists of setting up an individualized, intensive program (at least 20 hours per week) through the pleasure of play. The teacher follows the motivation and interests of the child, and it is the child who chooses the activities. Studies published in recent years tend to show that robots bring benefits to ASD children, particularly in the treatment of social interactions and in clinical settings. However, there is no scientific consensus on the generalized contribution and effect over time of these interventions. Moreover, a robotic solution controlled by a practitioner through a telepresence system allows for a better adaptability to the responses and desires of the children during the interventions. The investigators believe that such a solution would allow for better assessment of progress in the core skills of expressive communication and imitation and greater engagement during interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patient living in the Hérault department (France),
* Patient with a diagnosis of ASD confirmed by a psychiatrist or a psychologist and receiving current care according to the ESDM model in the MPEA Peyre Plantade child psychiatry service.

Exclusion Criteria:

* Patients

  * Failure to obtain written informed consent after a cooling-off period
  * Participating in another type of program other than ESDM
  * Not being affiliated to a French social security system or being a beneficiary of such a system
* Therapist

  * History of epilepsy for health professionals (therapists)

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-03-19 (Estimated); Study Completion 2025-09-19 (Estimated)

PRIMARY OUTCOMES:
Score of success on the selected task in the ESDM program | From phase A (baseline) to phase C (post-intervention) = 19 weeks
  Measure the success score for the selected task using the ESDM scoring grid. As soon as the child successfully completes one of the different learning stages, a success score is given to the task. This score will be maximum if all the learning stages of the task considered have been reached (Task 1 = 6 learning stages (maximum score =6); Tasks 2 and 3 = 7 stages (maximum score =7)). The ESDM scoring grid will be completed by the research therapists at the end of each session.

SECONDARY OUTCOMES:
Time of the child's viewing and movement of the head and body towards the robot (task 1: saying "hello") | During Phase B = 11 weeks
  Measurement of the viewing and movement times toward the robot, as well as the response time from the analysis of the videos made during the sessions using the Pepper robot.
  Data from the robot: - Video recording by camera of the sessions of the whole room (camera independent of the robot) - Video return by the camera installed on the robot - Audio feedback from the therapist, the robot and the child.

OTHER OUTCOMES:
Time of the child's viewing and movement of the head and body towards the therapist (task 1: saying "hello") | From phase A (baseline) to phase C (post-intervention) = 19 weeks
  Measurement of the viewing and movement times toward the therapist, as well as the response time from the analysis of the videos made during the sessions using the Pepper robot.
  Data from the robot: - Video recording by camera of the sessions of the whole room (camera independent of the robot) - Video return by the camera installed on the robot - Audio feedback from the therapist, the robot and the child.
Response time of the child after the presentation of the imitation exercise (task 2: action imitation) | From phase A (baseline) to phase C (post-intervention) = 19 weeks
  Measurement of the child's response time during the imitation exercise
Number of objects given to the robot (task 3 : give an object on verbal request) | From phase A (baseline) to phase C (post-intervention) = 19 weeks
  Measurement of the number of objects given out of the 5 requested (best score 5/5) in task 3.
Teleoperation success score for therapist (throught UX score) | Phase C (from week 5 to 15)
  Measurement of the success score (UX) of the teleoperation using the videos of the Pepper robot and according to the successful tasks to be performed during the session (the child and the second practitioner in the room can clearly hear the robot's instructions, the robot's gestures are fluid and is able to point to objects with the hand…). If the therapist was able to initiate each task, the score is 3/3.
Parent satisfaction score on current care | During phase A (to 4 weeks), Phase B (to 15 weeks), Phase C (to 19 weeks).
  Measurement of satisfaction score using a numerical satisfaction scale (EN). Parents will be asked about their current satisfaction with the care after each phase of the procedure. This will be rated on a scale of 0 to 10, (0 "I am not at all satisfied with the effectiveness of the proposed care" and 10 "I am totally satisfied with the care").
Professional satisfaction score on current care. | During phase A (to 4 weeks), Phase B (to 15 weeks), Phase C (to 19 weeks)
  Measurement of satisfaction score using a numerical satisfaction scale (EN). Professionals will be asked about their current satisfaction with the care after each phase of the procedure. This will be rated on a scale of 0 to 10, (0 "I am not at all satisfied with the effectiveness of the proposed care" and 10 "I am totally satisfied with the care").
Score of success in the ESDM tasks without teleoperation | During phase A (to 4 weeks), Phase C (from week 16 to 19
  This score (observe/total) will be maximum if all the learning stages of the task in question have been reached (Task 1 = 6 learning stages (maximum score =6); Tasks 2 and 3 = 7 stages (maximum score = 7)). This scoring will be done by therapist at the end of each intervention, after the current care.
Score of success in the ESDM tasks with teleoperation | During phase B (from week 5 to 15)
  This score (observe/total) will be maximum if all the learning stages of the task in question have been reached (Task 1 = 6 learning stages (maximum score =6); Tasks 2 and 3 = 7 stages (maximum score =7)).The robotics analyses will be performed by a robotic engineer of the LIRMM independent to the project.
Teleoperation usability score for therapist (throught UMUX score) | During phase A (to 4 weeks), Phase B (to 15 weeks), Phase C (to 19 weeks)
  A User Experience Questionnaire (UMUX) was administered at weeks 5, 10 and 15 to assess the quality and ease of use of the teleoperation system over time. The questionnaires are evaluated on a scale from 0 (minimum score) to 10 (maximum score). 0=Not at all satisfied 10= Totally satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital La Colombière - CHU de Montpellier, Montpellier, France

REFERENCES:
- [Derived] Fournier C, Michelon C, Granit V, Audoyer P, Bernardot A, Picot MC, Kheddar A, Baghdadli A. Pilot study protocol evaluating the impact of telerobotics interactions with autistic children during a Denver intervention on communication skills using single-case experimental design. BMJ Open. 2024 Nov 12;14(11):e084110. doi: 10.1136/bmjopen-2024-084110. PMID 39532363